CLINICAL TRIAL: NCT03167489
Title: Impact of Lifestyle Intervention Plus Emotion Regulation Group Intervention on Cardiovascular Risk Reduction in Women: A Pilot Study
Brief Title: Lifestyle Intervention Plus Emotion Regulation Group Intervention Impact on Women's Cardiovascular Risk Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Director of Linda Joy Pollin Cardiovascular Wellness Center for Women, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5579-HMO-CTIL
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Diseases; Lifestyle Risk Reduction
MeSH Terms: conditions — Cardiovascular Diseases; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: This pilot study includes a within subjects, delayed intervention design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle Plus Emotional Regulation (Experimental): The core intervention will last 5 months. Nutrition content: Mediterranean diet education, social support, self-regulation techniques, and environmental support. Physical activity content: education, guidance in starting a routine, and a walking program with pedometers, weekly physical activity tips and step goals. Emotion regulation content: based on Dialectical Behavior Therapy adapted to binge eating disorders and other ER sources, emphasizing identifying emotions, recognizing the causes of emotions, accepting and tolerating negative emotions, effective self-support and self-compassion, and the ability to manage situations that elicit negative emotions, as well as re-appraisal skills, which are identified as particularly influential on eating behaviors.
  Interventions: Behavioral: Lifestyle Plus Emotional Regulation

INTERVENTIONS:
Behavioral: Lifestyle Plus Emotional Regulation — Group intervention over 5 months, integrating the Mediterranean Diet into a lifestyle intervention and emotional regulation skills.

SUMMARY:
This pilot study aims to demonstrate that emotional regulation (ER) is a valuable supplement to a documented and effective group-based lifestyle intervention on cardiovascular disease risk reduction maintenance in a non-clinical population by assessing changes in this primary outcome: Mediterranean diet adherence and these secondary outcomes: average daily steps, METS per week, BMI, blood pressure, physical activity, LDL, HDL, Triglycerides, Hemoglobin A1c, Western Diet Score, ER skills, Healthy Heart Score and eating behavior. This study will include women aged 35-75 and the group intervention will be based on the gold standard Diabetes Prevention Study, integrating the Mediterranean Diet as well as emotional regulation skills based on dialectical behavior therapy. The core intervention will last 3 months with 2 booster sessions will be conducted over 1 month.

DETAILED DESCRIPTION:
Group lifestyle interventions (LI) have documented efficacy in improving cardiovascular disease (CVD) risk factors, however, many fail to demonstrate outcome maintenance. Existing LIs primarily focus on behavioral regulation, neglecting to address emotional regulation (ER). Difficulty with negative emotions often leads to unhealthy lifestyle recidivism, particularly in women, whereas acquiring ER skills have been found to improve healthy eating and is associated with increased physical activity. The effectiveness of ER as a healthy eating intervention has been documented in individuals with binge eating disorders and obese emotional eaters; however, it has never been utilized in a non-clinical population.

This pilot study aims to demonstrate that emotional regulation (ER) is a valuable supplement to a documented and effective group-based lifestyle intervention on cardiovascular disease risk reduction maintenance in a non-clinical population by assessing changes in this primary outcome: Mediterranean diet adherence and these secondary outcomes: average daily steps, METS per week, BMI, blood pressure, physical activity, LDL, HDL, Triglycerides, Hemoglobin A1c, Western Diet Score, ER skills, Healthy Heart Score and eating behavior. This study will include females and the group intervention will be based on the gold standard Diabetes Prevention Program, integrating the Mediterranean Diet as well as emotional regulation skills based on dialectical behavior therapy. The intervention will take place over 4 months: a weekly core intervention over 3 months time and 2 booster sessions over 1 month time.

Intervention:

Group sessions will focus on adherence to the Mediterranean Diet and increased physical activity. Nutrition content will include diet education, group counseling and social support, food interaction (tasting and cooking), behavioral self-regulation techniques (goal setting, self-monitoring, planning), conscious eating, creating healthy environmental support, and guidance tailored to the target audience. Physical activity will include education, motivation, guidance in starting a routine, and an experiential aerobic exercise class. Participants will be encouraged to exercise at least 150 minutes per week. Physical activity will also be integrated into sessions through a walking program, where participants receive a pedometer, weekly physical activity encouragement and tips, and create weekly step goals. Weekly steps will be tabulated by group leaders and assistants through pedometer measurement.

The emotion regulation skills modules will be modified from the Dialectical Behavior Therapy manual adapted to binge eating disorders (DBT-BED) and other ER sources. These modules will emphasize ER skills that include the ability to identify and label emotions, to recognize their causes and what maintains emotions, the ability to accept and tolerate negative emotions, the skills to provide effective self-support and self-compassion in distressing situations, and the ability to manage situations that elicit negative emotions, as well as re-appraisal skills, which are identified as particularly influential on eating behaviors.

Maintenance preparation sessions will address behavioral change maintenance, obstacle identification and coping skills. The booster session will provide an overview of the intervention and plans for continued outside-intervention support.

Data will be collected at baseline and 2 post intervention follow up points (after the first 4 months and 6 months following).

Control:

There will be a delayed treatment control for this pilot, wherein participants who enlist to the study will be asked complete baseline questionnaires at enlistment date, 4 months later (at the start of the intervention) and then, at the 2 post intervention data points.

ELIGIBILITY:
Inclusion Criteria:

- Women aged 35-75, willingness to commit to participation in the lifestyle intervention and follow-up.

Exclusion Criteria:

* Pregnancy, history of serious mental and physical illness, or other conditions that may impede or prohibit participation for the duration of the trial.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mediterranean Diet Adherence | 5 months after intervention initiation
  The Mediterranean Diet (MD) is an eating style that emphasizes the consumption of fruits, vegetables, legumes, and whole grains as well as fish, wine, olive oil, and nuts. MD adherence will be assessed through a self-report questionnaire based on the ATTICA Study, adapted to the Israeli diet (Panagiotakos, Chrysohoou, Pitsavos, and Stefanadis, 2005).

SECONDARY OUTCOMES:
Pedometer Steps | 5 months after intervention initiation
  Participants will be provided with a pedometer (Omron Model HJ-320) and will be encouraged to wear it throughout the program. Omron pedometers have been shown to demonstrate validity and reliability at various mounting positions in both healthy and overweight adults49. Measures will include average daily steps, as an objective measure of physical activity, and percentage change in steps, as an objective measure of change in physical activity level.
Body Mass Index | 5 months after intervention initiation
  Weight will be measured in kilograms using a standardized, calibrated scale and height will be measured using a standardized stadiometer. Weight loss in kilograms and percent weight loss will be calculated. BMI will be calculated by body weight /height2, and change in BMI will be calculated.
Blood Pressure | 5 months after intervention initiation
  Blood pressure will be measured using standard procedures with an electronic BP apparatus and the recorded measurement will be the average of 2 measurements taken in the seated position .
Hemoglobin A1c, plasma levels of HDL, LDL, triglycerides, and total cholesterol | 5 months after intervention initiation
  Hemoglobin A1c, plasma levels of HDL, LDL, triglycerides, and total cholesterol will be measured using capillary whole blood obtained on finger stick, through hospital and national health management organizations' laboratories.
Emotional Regulation Skills | 5 months after intervention initiation
  The Difficulties in Emotion Regulation Scale-16 (DERS-16) is a brief measure of emotion regulation difficulties. This scale demonstrates good internal consistency, test-retest reliability, as well as convergent and discriminant validity.
Eating Behavior | 5 months after intervention initiation
  The Dutch Eating Behavior Questionnaire (DEBQ) is a measure of Restrained, External, and Emotional eating. This questionnaire has good internal consistency and factorial validity as well as predictive validity for food consumption.
Healthy Heart Score | 5 months after intervention initiation
  The Healthy Heart Score is a lifestyle-based CVD prediction model that was developed using health data from 61,025 women in the Nurses' Health Study and 34,478 men in the Health Professionals Follow-up Study, who were free of chronic disease in 1986 and followed for CVD for up to 24 years. The Healthy Heart Score is based on the diet and lifestyle factors that include smoking, weight, exercise, and intake of alcohol, fruits and vegetables, whole grains, nuts, sugary beverages, and red and processed meat. On a prospective study, women with higher predicted CVD risk based on the Healthy Heart Score had an 18-fold higher risk of type 2 diabetes mellitus,5-fold higher risk of hypertension, and 3-fold higher risk of hypercholesterolemia during 20 years.
Binge Eating Behavior | 5 months after intervention initiation
  Binge eating behavior will assesses using items 13, 14 and 15 of the Eating Disorders Examination - Questionnaire (EDE-Q), as has been done previously by Goldfein and colleagues (Goldfein, 2005). The EDE-Q is the most reliable and valid instrument for eating disorder assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Donna R Zwas, MD, Principal Investigator — Hadassah University Medical Center
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stampfer MJ, Hu FB, Manson JE, Rimm EB, Willett WC. Primary prevention of coronary heart disease in women through diet and lifestyle. N Engl J Med. 2000 Jul 6;343(1):16-22. doi: 10.1056/NEJM200007063430103. PMID 10882764
- [Background] Roosen MA, Safer D, Adler S, Cebolla A, van Strien T. Group dialectical behavior therapy adapted for obese emotional eaters; a pilot study. Nutr Hosp. 2012 Jul-Aug;27(4):1141-7. doi: 10.3305/nh.2012.27.4.5843. PMID 23165554
- [Background] Neamah HH, Sebert Kuhlmann AK, Tabak RG. Effectiveness of Program Modification Strategies of the Diabetes Prevention Program: A Systematic Review. Diabetes Educ. 2016 Apr;42(2):153-65. doi: 10.1177/0145721716630386. Epub 2016 Feb 15. PMID 26879459
- [Background] Eckert M, Ebert DD, Lehr D, Sieland B, Jazaieri H, Berking M. Teachers' Emotion Regulation Skills Facilitate Implementation of Health-related Intentions. Am J Health Behav. 2015 Nov;39(6):874-81. doi: 10.5993/AJHB.39.6.15. PMID 26450555
- [Background] Macht M, Simons G. Emotions and eating in everyday life. Appetite. 2000 Aug;35(1):65-71. doi: 10.1006/appe.2000.0325. PMID 10896762
- [Background] Wallace LM, Masson PC, Safer DL, von Ranson KM. Change in emotion regulation during the course of treatment predicts binge abstinence in guided self-help dialectical behavior therapy for binge eating disorder. J Eat Disord. 2014 Dec 11;2(1):35. doi: 10.1186/s40337-014-0035-x. eCollection 2014. PMID 25516798